CLINICAL TRIAL: NCT01468558
Title: A Phase I Evaluation of the Effect of Ketoconazole on the Pharmacokinetics and Safety of Dihydroergotamine Mesylate (DHE) Delivered by Oral Inhalation (MAP0004) in Healthy Volunteers Compared to DHE Delivered Intravenously (DHE 45®)
Brief Title: Pharmacokinetics & Tolerability Study of MAP0004 Co-administered With Ketoconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: MAP Pharmaceuticals, Inc., a wholly owned subsidiary of Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAP0004-CL-P104
Record Dates: First submitted 2011-10-28; First posted 2011-11-09 (Estimated); Results first posted 2013-10-22 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: Drug Drug Interaction Study in Normal Healthy Volunteers
MeSH Terms: interventions — Dihydroergotamine; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Other): Subjects received MAP0004 on Day 1 of Visit 2, Ketoconazole on Days 3 through 6 of Visit 2, and MAP0004 again on Day 6 of Visit 2. Subjects then returned for Visit 3, 7-11 days from the end of Visit 2. At Visit 3 subjects received 1.0 mg IV DHE (Intravenous Dihydroergotamine Mesylate).
  Interventions: Drug: MAP0004; Drug: IV DHE; Drug: Ketoconazole

INTERVENTIONS:
Drug: MAP0004 — MAP0004 1.0mg via inhalation on Day 1 and Day 6 of Visit 2
Drug: IV DHE — IV DHE (Intravenous Dihydroergotamine Mesylate) administered at Visit 3
  Other Names: D.H.E.45®
Drug: Ketoconazole — Ketoconazole 400 mg administered once a day on days 3-6 of Visit 2
  Other Names: Nizoral®

SUMMARY:
Compare the DHE pharmacokinetic profiles observed following administration of:

1. MAP0004 (oral inhalation DHE)
2. MAP0004 co-administered with oral Ketoconazole
3. Intravenous (IV) DHE (D.H.E.45®, the approved reference therapy)

Compare the tolerability of MAP0004, IV DHE, and MAP0004 with co-administration of Ketoconazole.

ELIGIBILITY:
Major Inclusion Criteria:

* Able to provide written Informed Consent
* Male or Female subjects 18 to 45 years old
* Female subjects who are practicing adequate contraception or who are sterile
* Stable cardiac status
* Normal rhythm or arrhythmia deemed clinically insignificant on ECG

Exclusion Criteria:

* Contraindication to dihydroergotamine mesylate (DHE)
* Use of any excluded concomitant medications within the 10 days prior to Visit 1
* History of hemiplegic or basilar migraine
* Participation in another investigational trial during the 12 weeks prior to Visit 1 or during this trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Simbec Research Limited, Merthyr Tydfil, Merthyr Tydfil, United Kingdom

REFERENCES:
- [Derived] Kellerman D, Kori S, Forst A, Chang J, Febbraro S, Wutann L, Thomas T, Taylor G, Dodick D. Lack of drug interaction between the migraine drug MAP0004 (orally inhaled dihydroergotamine) and a CYP3A4 inhibitor in humans. Cephalalgia. 2012 Jan;32(2):150-8. doi: 10.1177/0333102411432299. Epub 2011 Dec 15. PMID 22174351

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects received MAP0004 on Day 1 of Visit 2, Ketoconazole on Days 3 through 6 of Visit 2, and MAP0004 again on Day 6 of Visit 2. Subjects then returned for Visit 3, 7-11 days from the end of Visit 2. At Visit 3 subjects received 1.0 mg Intravenous (IV) Dihydroergotamine Mesylate (DHE).
Groups:
- Overall Study: Subjects first received MAP0004 1.0mg via oral inhalation followed by 48 hours of PK sampling, they then received Ketoconazole (400mg once a day for 4 days) followed by MAP0004 1.0mg and another 48 hours of PK sampling. After a 7-11 day washout, subjects returned to the clinic to receive 1.0mg IV DHE and 48 hours of PK sampling.
Period: Overall Study
Arm/Group | Overall Study
Started | 24
Completed | 22
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All subjects that were enrolled in the study.
Arm/Group | Overall Study
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.58 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Dihydroergotamine After MAP0004, MAP0004 Co-administered With Ketoconazole, and IV DHE Administration
Description: The maximum concentration (Cmax) is the highest concentration of a drug measured in the plasma. Plasma is the clear portion of the blood. The Cmax of Dihydroergotamine is reported in picograms per milliliter (pg/ml).
Time Frame: 48 hours
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Geometric Mean (Standard Deviation); unit: pg/ml
Groups:
- MAP0004 1.0mg: MAP0004 1.0mg via inhalation on Day 1 of Visit 2.
- MAP0004 1.0mg + Ketoconazole: Ketoconazole 400mg once a day on Days 3-6 of Visit 2 and MAP0004 1.0mg via inhalation on Day 6 of Visit 2.
- IV DHE 1.0mg: IV DHE 1.0mg on Day 1 of Visit 3.
Arm/Group | MAP0004 1.0mg | MAP0004 1.0mg + Ketoconazole | IV DHE 1.0mg
Number analyzed (Participants) | 21 | 23 | 20
pg/ml | 2582.507 (1137.829) | 2495.100 (1130.850) | 27771.234 (36191.528)

2. Primary Outcome: AUC(0-48) of Dihydroergotamine After MAP0004, MAP0004 Co-administered With Ketoconazole, and IV DHE Administration
Description: The AUC(0-48) is the area under the plot of plasma concentration of drug against time after drug administration. Dihydroergotamine AUC(0-48) is reported in picograms times hour per milliliter (pg*h/ml).
Time Frame: 48 hours
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Geometric Mean (Standard Deviation); unit: pg*h/ml
Arm/Group | MAP0004 1.0mg | MAP0004 1.0mg + Ketoconazole | IV DHE 1.0mg
Number analyzed (Participants) | 23 | 23 | 20
pg*h/ml | 3484.725 (1221.423) | 4070.611 (1628.973) | 9229.171 (3130.093)

ADVERSE EVENTS:
Description: All 24 subjects who received MAP0004 alone, 24 subjects who received MAP0004 with ketoconazole, and 22 subjects who received IV DHE are included in the adverse event analysis. Adverse events are presented by treatment arm, not necessarily by individual treatment (intervention) received.
Arm/Group | MAP0004 1.0mg | MAP0004 1.0mg + Ketoconazole | IV DHE 1.0mg
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 6/24 | 7/24 | 11/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MAP0004 1.0mg (N=24) | MAP0004 1.0mg + Ketoconazole (N=24) | IV DHE 1.0mg (N=22)
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 11
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Dizziness (Nervous system disorders) | 1 | 1 | 4
Headache (Nervous system disorders) | 6 | 7 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hot flush (Vascular disorders) | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.